CLINICAL TRIAL: NCT04710797
Title: A Prospective Randomized Multicentre Trial for Lymphadenectomy in Early-stage Ovarian Cancer
Brief Title: Lymphadenectomy in Early Ovarian Cancer
Acronym: LOVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jihong Liu, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-FXY-405
Record Dates: First submitted 2021-01-11; First posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Ovarian Cancer; Lymphadenectomy
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: comprehensive staging surgery with or without lymphadenectomy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Lymphadenectomy (Experimental): Comprehensive staging surgery with no Lymphadenectomy
  Interventions: Procedure: Comprehensive staging surgery with no Lymphadenectomy
- Lymphadenectomy (Active Comparator): Completion staging surgery including systematic pelvic and para-aortic lymphadenectomy
  Interventions: Procedure: Completion staging surgery including systematic pelvic and para-aortic lymphadenectomy

INTERVENTIONS:
Procedure: Completion staging surgery including systematic pelvic and para-aortic lymphadenectomy — * open or minimally invasive surgical approach
  * cytologic examinations
  * All peritoneal surfaces should be visualized, and any peritoneal suspicious for metastasis should be selectively excised or biopsied
  * BSO and hysterectomy
  * For selected patients desiring to preserve fertility, USO or BSO with uterine preservation may be considered
  * Omentectomy
  * Para-aortic lymph node dissection should be performed by stripping the nodal tissue from the vena cava and the aorta bilaterally to at least the level of the inferior mesenteric artery and preferably to the level of the renal vessels
  * The preferred method of dissecting pelvic lymph nodes is bilateral removal of lymph nodes overlying and anterolateral to the common iliac vessel, overlying and medial to the external iliac vessel, overlying and medial to the hypogastric vessels, and from the obturator fossa at a minimum anterior to the obturator nerve
  Arms: Lymphadenectomy
Procedure: Comprehensive staging surgery with no Lymphadenectomy — * open or minimally invasive surgical approach
  * cytologic examinations
  * All peritoneal surfaces should be visualized, and any peritoneal suspicious for metastasis should be selectively excised or biopsied
  * BSO and hysterectomy
  * For selected patients desiring to preserve fertility, USO or BSO with uterine preservation may be considered
  * Omentectomy
  * In open approach surgery, exploring the pelvic and Para-aortic lymph node with hand. In minimally invasive surgery, the peritoneal above the pelvic and Para-aortic lymph node area should be open and visualized.Biopsy and frozen section of the suspicious lymph nodes
  Arms: No Lymphadenectomy

SUMMARY:
To assess the impact of comprehensive staging surgery with no lymphadenectomy on survival and quality of life in patients with early-stage ovarian cancer.

DETAILED DESCRIPTION:
OBJECTIVES: Compare the efficacy and safety in patients with International Federation of Gynecology and Obstetrics (FIGO) stage IA -IIA epithelial ovarian cancer, undergo completion staging surgery including systematic pelvic and para-aortic lymphadenectomy versus comprehensive staging surgery without lymphadenectomy.

OUTLINE: This is a randomized phase III multicenter study. Patients will receive comprehensive staging surgery without Lymphadenectomy or completion staging surgery including systematic pelvic and para-aortic lymphadenectomy, and the adjuvant chemotherapy will accord to National Comprehensive Cancer Network (NCCN) guidelines. Patients are followed up every 3 months within the first 2 years, and then every 6 months.

PROJECTED ACCRUAL: A total of 656 patients will be recruited for this study within 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18 years to 70 years.
2. Primary diagnosis of epithelial ovarian cancer FIGO stage IA-IIA ( recevive no prior treatment or receive incomplete initial surgery)，with indications of adjuvant chemotherapy：①High-grade serous carcinoma; ②Grade 3 endometrioid carcinoma; ③Clear cell carcinoma; ④Grade 2 endometrioid carcinoma with capsule ruptured or pelvic tissues extension ⑤Low-grade serous carcinoma、Grade 1 endometrioid carcinoma and Mucinous carcinoma of the ovary with pelvic tissues extension.
3. Patients who have given their signed and written informed consent.
4. Good performance status (ECOG 0/1).

Exclusion Criteria:

1. Non epithelial ovarian malignancies and borderline tumors.
2. Suspicious lymph nodes at preoperative radiological evaluation.
3. Intraoperative clinically suspicious lymph nodes (bulky nodes).
4. Secondary invasive neoplasms in the last 5 years (except synchronal endometrial carcinoma FIGO IA G1/2, non melanoma skin cancer, breast cancer T1 N0 M0 G1/2) or with any signs of relapse or activity.
5. Prior chemotherapy for ovarian cancer or abdominal/pelvic radiotherapy.
6. Diseases of the lymph system (including lymph edema of unknown origin).
7. Prior retroperitoneal lymph node dissection (systematic or sampling).
8. Any other concurrent medical conditions contraindicating surgery.
9. Pregnancy.
10. Any reasons interfering with giving of informed consent , abiding by protocol, or regular follow-up.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 656 (Estimated)
Dates: Start 2021-01-31 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS(Progression-free survival) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  From date of randomization until the date of first documented progression or date of death from any cause, whichever came first

SECONDARY OUTCOMES:
OS(Overall Survival) | From date of randomization until the date of death from any cause or date of last follow up, up to 100 mons
  From date of randomization until the date of death from any cause or date of last follow up, whichever came first
Recurrence rate of lymph node | 3 years
  The recurrence rate in the retroperitoneal lymph nodes after primary surgery
QoL(Quality of life) | Baseline, 6 months and 1 year after surgery
  Quality of life before surgery, and at 6 months and 1 year after surgery in both groups will be evaluated using European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire
Postoperative complications | 3 years
  The difference of the rate of Postoperative complications between two groups

CONTACTS AND LOCATIONS:
Overall Officials: Jihong Liu, Ph.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Department of Gynecologic Oncology, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Deng T, Liu K, Chen L, Chen X, Li HW, Guo H, Zhang H, Xiang L, Feng X, Wang X, Ngan HY, Zhao J, Zou D, Liu Q, Liu J. A prospective randomized multicenter trial for lymphadenectomy in early-stage ovarian cancer: LOVE study. J Gynecol Oncol. 2023 May;34(3):e52. doi: 10.3802/jgo.2023.34.e52. Epub 2023 Apr 10. PMID 37116952